CLINICAL TRIAL: NCT03466294
Title: Azacitidine and Venetoclax (ABT-199) as Induction Therapy With Venetoclax Maintenance in Previously Untreated Elderly Patients With Acute Myeloid Leukemia (AML)
Brief Title: Azacitidine and Venetoclax as Induction Therapy With Venetoclax Maintenance in the Elderly With AML
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-7821.cc
Record Dates: First submitted 2018-03-02; First posted 2018-03-15 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Acute Myeloid Leukemia
Keywords: Azacitidine; Venetoclax; AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Azacitidine; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Azacitidine and Venetoclax (Experimental): On day 1 of cycle 1, Azacitidine 75 mg/m2 will be given by injection or infusion, and will continue for 7 days. Azacitidine doses will be given in subsequent cycles for patients who do not achieve response. Venetoclax will be administered orally once daily on days 2 through 28 in cycle 1. Beginning with cycle 2, and each subsequent cycle, venetoclax will be administered Days 1 through 28.
  Interventions: Drug: Azacitidine and Venetoclax

INTERVENTIONS:
Drug: Azacitidine and Venetoclax — Azacitidine will be given at dose of 75mg/m2 in Cycle 1 days 1-7; repeat in cycle 2 and 3 if no response. Starting on day 2 of cycle 1, venetoclax will be administered orally with doses increased to a target dose of 600 mg (administer 100 mg on day 2, 200 mg on day 3, 400 mg on day 4 and 600 mg on day 5), then 600 mg daily.

SUMMARY:
This study is being done to determine if treatment with azacitidine and venetoclax is effective treatment for elderly patients with acute myeloid leukemia (AML) who have not received previous treatment. Azacitidine and venetoclax will be given as induction treatment followed by venetoclax maintenance treatment for patients who respond to the induction treatment.

DETAILED DESCRIPTION:
This is a phase 2 study for elderly patients who have not received previous treatment for acute myeloid leukemia (AML). Up to 42 patients will be enrolled. All patients will be treated with azacitidine and venetoclax until a minimal residual disease (MRD) negative response is achieved. Once patients achieve a MRD negative composite response, azacitidine will be discontinued and venetoclax dose will be decreased to "maintenance" dose.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must have confirmation of non-APL AML by WHO criteria and be ineligible or unwilling to undergo treatment with a standard cytarabine and anthracycline induction regimen due to co-morbidities or other factors
2. Subject must have received no prior treatment for AML; hydroxyurea is not considered a treatment and is allowed
3. Subject must be ≥ 60 years of age
4. Subject must have a projected life expectancy of at least 12 weeks
5. Subject must have an Eastern Cooperative Oncology Group (ECOG) Performance status of ≤2
6. Subject must have adequate renal function as demonstrated by a calculated creatinine clearance ≥ 30 mL/min; determined via urine collection for 24-hour creatinine clearance or by the Cockcroft Gault formula
7. Subject must have adequate liver function as demonstrated by:

   * aspartate aminotransferase (AST) ≤ 3.0 × ULN*
   * alanine aminotransferase (ALT) ≤ 3.0 × ULN*
   * bilirubin ≤ 3.0 × ULN, unless due to Gilbert's syndrome*

     * Unless considered due to leukemic organ involvement
8. Non-sterile male subjects must use contraceptive methods with partner(s) prior to beginning study drug administration and continuing up to 90 days after the last dose of study drug. Male subjects must agree to refrain from sperm donation from initial study drug administration until 90 days after the last dose of study drug.
9. Female subjects must be either:

   * Postmenopausal; defined as Age > 55 years with no menses for 12 or more months without an alternative medical cause; OR
   * Permanently surgically sterile (bilateral oophorectomy, bilateral salpingectomy or hysterectomy)
10. Subject must voluntarily sign and date an informed consent, approved by an Institutional Review Board (IRB), prior to the initiation of any screening or study-specific procedures.

Exclusion Criteria:

1. Subject has received treatment with a hypomethylating agent and/or other chemotherapeutic agent either conventional or experimental for myelodysplastic syndrome (MDS) or AML
2. Subject has acute promyelocytic leukemia
3. Subject has known active CNS involvement from AML
4. Subject is known to be positive for HIV. HIV testing is not required
5. Subject is known to be positive for hepatitis B or C infection with the exception of those with an undetectable viral load. Hepatitis B or C testing is not required and subjects with serologic evidence of prior vaccination to HBV (i.e., HBs Ag, anti-HBs+ and anti-HBc-) may participate
6. Subject has received anticancer therapies including chemotherapy, radiotherapy or other investigational therapy, including targeted small molecule agents within 5 half-lives prior to first dose of study drug
7. Subject has received biologic agents (e.g. monoclonal antibodies) for anti-neoplastic intent within 30 days prior to first dose of study drug
8. Subject has received the following within 7 days prior to the first dose of the study drug:

   * Steroid therapy for anti-neoplastic intent;
   * Strong and Moderate CYP3A inhibitors (see Appendix A for examples)
   * Strong and Moderate CYP3A inducers (see Appendix A for examples)
9. Subject has consumed grapefruit, grapefruit products, Seville oranges (including marmalade containing Seville oranges) or Star fruit within 3 days prior to the initiation of study treatment
10. Subject has any history of clinically significant condition(s) that in the opinion of the investigator would adversely affect his/her participating in this study including, but not limited to:

    * New York Heart Association heart failure > class 2
    * Renal, neurologic, psychiatric, endocrinologic, metabolic, immunologic, hepatic, cardiovascular disease, or bleeding disorder independent of leukemia
11. Subject has a malabsorption syndrome or other condition that precludes enteral route of administration
12. Subject exhibits evidence of uncontrolled systemic infection requiring therapy (viral, bacterial or fungal)
13. Subject has a history of other malignancies prior to study entry, with the exception of:

    * Adequately treated in situ carcinoma of the breast or cervix uteri
    * Basal cell carcinoma of the skin or localized squamous cell carcinoma of the skin
    * Prostate cancer with no plans for therapy of any kind
    * Previous malignancy confined and surgically resected (or treated with other modalities) with curative intent
14. Subject has a white blood cell count > 25 × 109/L. Note: hydroxyurea is permitted to meet this criteria
15. Any subject who is a candidate for intensive induction therapy and agrees to receive this therapy

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2018-05-15 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Duration of response to azacitidine and venetoclax treatment | From the first day a response is documented to the first day of disease progression
  Determine how long responses last in patients treated with azacitidine and venetoclax followed by venetoclax maintenance treatment

SECONDARY OUTCOMES:
Frequency of Minimal Residual Disease (MRD) negative composite responses within the "induction phase" of azacitidine and venetoclax | From Day 28, the first day a response is documented to end of cycle bone marrow biopsies, through 5 years
  The number of patients who achieve an MRD negative composite response
The time needed to achieve an MRD negative composite response | From first dose of treatment to first day response is documented by bone marrow biopsy
  The median number of days that have elapsed leading to an MRD negative composite response
The one-year overall survival (OS) of older, newly diagnosed AML patients treated with "induction phase" of azacitidine with venetoclax followed by a maintenance Phase of venetoclax alone. | From date of study enrollment to one year after enrollment
  The number of patients who survive to one year after date of study enrollment
Hematologic Toxicity as defined by the 2017 ELN AML Recommendations | From the day venetoclax with azacitidine is administered to the end of maintenance venetoclax alone, up to one year
  Hematologic toxicities will be measured by incidence of febrile neutropenia, ≥ grade 2 bleeding complications and number of transfusions received

CONTACTS AND LOCATIONS:
Overall Officials: Dan Pollyea, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shallis RM, Podoltsev NA. Maintenance therapy for acute myeloid leukemia: sustaining the pursuit for sustained remission. Curr Opin Hematol. 2021 Mar 1;28(2):110-121. doi: 10.1097/MOH.0000000000000637. PMID 33394722